CLINICAL TRIAL: NCT01880775
Title: The Comparison of the Discharge Conditions and Efficacy of Spinal Anesthesia With Heavy Prilocaine-Fentanyl and Heavy Bupivacaine-Fentanyl in Outpatient Minor Perianal Surgery
Brief Title: Discharge Conditions of Spinal Anesthesia With Heavy Prilocaine-Fentanyl and Heavy Bupivacaine-Fentanyl
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozden Gorgoz Kaban, Medical Doctor Trainee in Anesthesiology and Reanimation, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: OKabanPrilocain
Record Dates: First submitted 2012-03-12; First posted 2013-06-19 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2012-03

CONDITIONS: Hemorrhoid; Peri Anal Fistula
MeSH Terms: conditions — Hemorrhoids | interventions — Prilocaine; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prilocaine heavy 2%& fentanyl (Experimental): prilocaine heavy 2% 30 mg and fentanyl 20 micgr ampoule intrathecal
  Interventions: Drug: Prilocaine
- bupivacaine heavy 0.5% & fentanyl (Active Comparator): bupivacaine heavy 0.5% 7.5 mg and fentanyl 20 micg ampoule intrathecal
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Prilocaine — experimental
  Other Names: prilothecal; citanest
  Arms: prilocaine heavy 2%& fentanyl
Drug: Bupivacaine — marcaine heavy 0.5% 7.5 mg intrathecal
  Other Names: marcaine heavy 0.5%
  Arms: bupivacaine heavy 0.5% & fentanyl

SUMMARY:
In this prospective randomized study the investigators aimed to investigate difference of the duration of spinal anesthesia, discharge times and efficacy between low dose heavy Prilocaine-Fentanyl and heavy Bupivacaine-Fentanyl in outpatient minor anal surgery.

DETAILED DESCRIPTION:
ASA status I-III patients will be recruited. Patients will be randomized in two groups. Group B will be received 1.5 ml heavy bupivacaine+ 20 mic fentanyl+ 0.15 ml and Group P will be received 1,5 ml heavy prilocaine+20 mic fentanyl in the same volume.Patients will be monitored with electrocardiography, peripheral oxygen saturation(sPO2) and non invasive blood pressure (Drager Infinity Delta; 16 Electronics Avenue, Danvers, MA 01923 USA). After inserting a 20 G intravenous line the patients will be hydrated with 10 ml/kg 0.9 % saline.

Preoperative systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP), heart rate (HR) and Spo2 will be measured and recorded.

Spinal anesthesia will be commenced in the sitting position with a 25 G Quincke needle, with the midline approach. After observing free flow of cerebrospinal fluid the prepared study drug will be injected in 15 seconds. The patients will be placed supine after waiting 2 minute in the sitting position. Supplemental oxygen via nasal cannula will be provided.

Fentanyl and midazolam will be used for rescue analgesia and sedation and recorded.

Sensorial block will be assessed with pinprick test with 2 minute intervals until the maximum block achieves and with 15 minute intervals until the block was regresses to S3 dermatome. Motor block will be assessed with the Bromage score when the block reached the maximum level. Patients will be transferred to postoperative care unit (PACU) at he end of surgery.

Pain will be assessed on a 10 point visual analog scale (VAS)(0= no pain, 10= worst pain ever). Postoperative analgesia will be provided with 2 mg.kg-1 tramadol or 15 mg.kg-1 paracetamol when the VAS score is ≥3 time of first analgesic request will be recorded.

Hypotension (≥20% reduced from baseline values) will be treated with ephedrine or iv fluid boluses), bradycardia (HR<45 beat min-1 was treated with atropine) was recorded.

The patients will be asked whether to void before surgery. Bladder volume will be assessed with ultrasonography. Patients with residual bladder volumes ≥400 ml will be placed an urine catheter. Time to first urinate will be recorded.

Patients will be assessed for transient neurologic symptoms(pain in the buttocks and legs)(TNS) and satisfaction after surgery.

TNS will be evaluated with daily telephone calls. Patient satisfaction will be evaluated with global satisfaction scale (1= bad, 2=not satisfied, 3=have no idea, 4=satisfied, 5=very satisfied) Parameters to record; time of entering operation room, duration of surgery, time of intrathecal injection, onset of sensorial block(block at L1), time to reach maximum block level, maximum block level, first analgesic ingestion time, PACU duration, two segment regression, time to L1 regression, time to S3 regression, time to it without help, time to stand up without help, time to walk without help, discharge time, time to first void. TNS, patient satisfaction score.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I-III

Exclusion Criteria:

* Patients with contraindications for spinal anesthesia,
* hypersensitivity to study drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Sensory block regression at S3 (time, minute) | postoperative 30. minute
  spinal anesthesia

SECONDARY OUTCOMES:
discharge time (minute) | postoperative 2 hour
  spinal anesthesia

OTHER OUTCOMES:
Maximum block height | Intraoperative 30 minutes
  Maximum spread of the sensorial block
Motor block | Intraoperative 30 minutes and postoperative first hour
  Bromage scale will be used 0: no motor block, 1: hip blocked, 2: hip and knee blocked, 3: hip, knee and ankle blocked
Regression of motor block | Postoperative second hour
  Bromage scale will be used 0: no motor block, 1: hip blocked, 2: hip and knee blocked, 3: hip, knee and ankle blocked
Time to L1 block | Intraoperative 5 minutes
  Loss of sensation to pin prick
Time to T10 block | Introperative 10 minute
  loss of sensation to pinprick

CONTACTS AND LOCATIONS:
Overall Officials: Taylan Akkaya, Assoc Prof., Study Director — Ministry of Health
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Camponovo C, Fanelli A, Ghisi D, Cristina D, Fanelli G. A prospective, double-blinded, randomized, clinical trial comparing the efficacy of 40 mg and 60 mg hyperbaric 2% prilocaine versus 60 mg plain 2% prilocaine for intrathecal anesthesia in ambulatory surgery. Anesth Analg. 2010 Aug;111(2):568-72. doi: 10.1213/ANE.0b013e3181e30bb8. Epub 2010 Jun 7. PMID 20529983
- [Background] Black AS, Newcombe GN, Plummer JL, McLeod DH, Martin DK. Spinal anaesthesia for ambulatory arthroscopic surgery of the knee: a comparison of low-dose prilocaine and fentanyl with bupivacaine and fentanyl. Br J Anaesth. 2011 Feb;106(2):183-8. doi: 10.1093/bja/aeq272. Epub 2010 Oct 14. PMID 20947591
- [Background] Ostgaard G, Hallaraker O, Ulveseth OK, Flaatten H. A randomised study of lidocaine and prilocaine for spinal anaesthesia. Acta Anaesthesiol Scand. 2000 Apr;44(4):436-40. doi: 10.1034/j.1399-6576.2000.440413.x. PMID 10757577